CLINICAL TRIAL: NCT02028494
Title: Evaluation of Response to Two Schedules of Capecitabine in Patients With Metastatic Breast Cancer
Acronym: CAP7/7
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Latin American & Caribbean Society of Medical Oncology (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLACOM Cap 7/7
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Capecitabine 2,000 mg (flat dose) (Experimental): Arm A: Capecitabine 2,000 mg (flat dose), orally, twice daily for 7 days followed by a 7 day rest (7-7) (4-week cycle length ).
  Interventions: Drug: Capecitabine
- Arm B: Capecitabine 1,000 mg/m2 twice daily for 14 day (Active Comparator): Arm B: Capecitabine 1,000 mg/m2, orally, twice daily for 14 days followed by a 7 day rest (14-7) (3-week cycle length ). The control arm dose of capecitabine has been reduced from the US Food and Drug Administration approved dose of 1,250 mg/m2, orally, twice daily due to common clinical practice.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Two dosages comparison
  Other Names: Xeloda

SUMMARY:
The purpose of this study is to compare the efficacy of a novel schedule of an oral anticancer drug, capecitabine, in patients with metastatic breast cancer.

Mathematical models have predicted that 7 days of capecitabine followed by 7 days of rest is an optimal dosing schedule for this drug and previous studies done al Memorial Sloan Kettering Cancer Center support the tolerability of this scheme.

This definitive, randomized trial comparing the efficacy of the new dosage with the conventional dosing schedule in patients with metastatic breast cancer is necessary and we hypothesize it will be superior in terms of efficacy.

Dosing schedules based on mathematical predictions for optimal drug delivery based on efficacy rather than toxicity could facilitate more rapid and economical drug development. This trial is a proof of principle trial of the highest priority.

ELIGIBILITY:
Inclusion Criteria:

* 1 Subject Inclusion Criteria

  * Informed consent has been obtained.
  * Metastatic breast cancer.
  * Measurable or non-measurable disease per RECIST criteria.
  * Pathologic confirmation of breast cancer.
  * No limit to the number of prior chemotherapy regimens permitted for metastatic disease.
  * At least 3 weeks since prior chemotherapy. Patients should have recovered from all acute toxicity from such therapy (excluding alopecia).
  * Age ≥18.
  * ECOG 0-2
  * Absolute Neutrophil Count (ANC )≥1.0; hemoglobin ≥9, platelets

    ≥75.000
  * AST, ALT and Alkaline phosphatase <2.5x upper limit of normal (or <5x upper limit of normal in the case of liver metastases). Total bilirubin <1.5x upper limit of normal.
  * Estimated creatinine clearance >50ml/min.
  * If female of childbearing potential, pregnancy test is negative and the patient agrees to use an effective method to avoid pregnancy during the study.

Exclusion Criteria:

* HER2 over-expression and/or amplification as determined by immunohistochemistry (3+) or FISH (>2.0).

  * No prior fluoropyrimidine in the metastatic setting. Adjuvant fluoropyrimidine is permitted if >12 months have elapsed since treatment.
  * No restriction for prior hormonal therapy.
  * GI malabsorption syndrome which could impair oral drug absorption.
  * Concurrent use of warfarin is discouraged as drug interactions may make management of INR more difficult.
  * Central nervous system metastases are permitted if previously treated or clinically stable for at least 3 months.
  * Pregnant or nursing patients.
  * Life expectancy <3 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2013-08; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival (PFS) | 24 month
  The primary endpoint of this study is PFS, defined as the time from treatment start to progression or last date of follow-up. PFS will be estimated using Kaplan-Meier methods. This will be an intention to treat analysis. The Log-rank test will be used to test whether PFS is different for the two capecitabine schedules. It is hypothesized that the 7-7 schedule of capecitabine will have superior efficacy.

SECONDARY OUTCOMES:
Number of participants with toxicity. | 24 month
  Secondary Objectives:
  * To assess and compare tolerability of the two capecitabine schedules in terms of selected hematologic and non-hematologic toxicities.
  * To compare the rates of grade 3 or greater diarrhea, nausea and vomiting between the two schedules.
Number of patients with treatment delays. | 24 month
Number of patients with dose reduction. | 24 month
Number of patients with study withdrawal. | 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Cazap, MD,PhD, Study Chair — Latin American & Caribbean Society of Medical Oncology; Tiffany Traina, MD, Study Chair — MSKCC
Locations (1):
- SLACOM, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided